CLINICAL TRIAL: NCT01317979
Title: Asian Diabetes Surgery Study:A Multi-institutes Prospective Study Clinical Predictor for the Successful Treatment of Type 2 Diabetes After Metabolic Surgery
Brief Title: Asian Diabetes Surgery Study (ADSS): Clinical Predictor for the Success of Metabolic Surgery
Acronym: ADSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Min-Sheng General Hospital IRB, Min-Sheng General Hospital IRB
Other Study IDs: MSIRB2011003
Record Dates: First submitted 2011-03-02; First posted 2011-03-18 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Disease; Endocrine System Disease; Diabetes Mellitus
MeSH Terms: conditions — Disease; Endocrine System Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum stored at a -85 ℃ refrigerator
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes group I: metabolic surgery, laparoscopicly

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a serious health problem that has increased dramatically worldwide due to the high and increasing prevalence of obesity. Medical management of T2DM is of limited success. Because not well controlled T2DM patients are in high risk of blindness, cardiovascular accident and end staged disease, T2DM has become a major health burden for society. Recent data on the relative effectiveness of gastrointestinal metabolic surgery played as bariatric surgery in the remission of T2DM, suggests that it may be significantly more effective than current medical treatment. In considering that less than half of the T2DM patients can achieve satisfactory treatment goal under current medical treatment, gastrointestinal metabolic surgery shall play an important role in T2DM treatment in the future. However, the indication for metabolic surgery and clinical predictors of success are not clear now. These clinical predictors can help us to choose appropriate not-well controlled T2DM patients to receive metabolic surgery and reduce dverse health outcomes in those patients.

DETAILED DESCRIPTION:
The present research proposal is designed to assess the clinical predictors of success in T2DM patients who receive metabolic surgery for the treatment of their diabetes. This study will recruit 200 obese T2DM patients who receive gastrointestinal metabolic surgery in our center and follow up them for one year. The Inclusion criteria are those with T2DM more than 6 months, age between 18 to 65 and HbA1C > 8%. All the pre-operative clinical parameters will be collected prospectively, including C-peptide and stimulated C-peptide. The genetic polymorphism of these patients will also be analyzed and collected. The success of T2DM remission will be assessed at 12 months after metabolic surgery will be composite endpoint of CVD risk factor resolution; specifically, the proportion of patients with HbA1c < 6.5%. The clinical predictors will be analyzed by uni-vriate and muti-variate analysis. In the first year project, we will included 100 patients and will include another 100 patients at the second year. This project will apply for the budget of 1st year.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65.
* Type 2 DM > 6 months, HbA1C>8.0% under treatment
* Body mass index >25 kg/m2
* could follow up

Exclusion Criteria:

* Age <18 or >65
* HbA1C < 7%
* BMI < 25 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Age between 18 to 65.
  2. Type 2 DM > 6 months, HbA1C>7.0% under treatment
  3. Body mass index >25 kg/m2
  4. could follow up
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-03 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Juin Tsou, university, Principal Investigator — Metabolic surgery center,Minsheng general hospital
Locations (2):
- Taiwan (2):
  - Min sheng general hospital, Taoyuan
  - MinSheng Genral Hospital, Taoyuan District